CLINICAL TRIAL: NCT02036801
Title: The Specific Elastance in ARDS Patients. Connections Between Volutrauma and Barotrauma - A Pediatric Study
Brief Title: The Specific Elastance in ARDS Patients: a Pediatric Study
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: policlinico-10
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Pediatric ARDS
Keywords: ARDS; Lung; Specific Elastance; Pediatric patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ARDS: Patients with ARDS (according to the Berlin Definition criteria) in mechanical ventilation
  Interventions: Other: Lung specific elastance
- Healthy control: Patients with healthy lung supported with mechanical ventilation for clinical purposes
  Interventions: Other: Lung specific elastance

INTERVENTIONS:
Other: Lung specific elastance — Measurement of lung specific elastance and lung mechanical characteristics at different PEEP levels and tidal volumes

SUMMARY:
Aim of this study is to assess lung specific elastance in a population of pediatric patients with Acute Respiratory Distress Syndrome (ARDS) treated with mechanical ventilation, and in a pediatric population of ICU patients with healthy lung which are treated with mechanical ventilation for other clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* ARDS (Berlin Definition Criteria) or mechanical ventilation in healthy lungs

Exclusion Criteria:

* Hemodynamic instability
* Lung diseases other than ARDS
* Parental refuse

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ARDS pediatric patients in mechanical ventilation or patients with healthy lung treated with mechanical ventilation for clinical purposes
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Specific elastance of the lung | 10 minutes from the start of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCC Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Derived] Chiumello D, Chidini G, Calderini E, Colombo A, Crimella F, Brioni M. Respiratory mechanics and lung stress/strain in children with acute respiratory distress syndrome. Ann Intensive Care. 2016 Dec;6(1):11. doi: 10.1186/s13613-016-0113-0. Epub 2016 Feb 5. PMID 26847436